CLINICAL TRIAL: NCT06031142
Title: Flexible Wearable Device for Continuous Fetal Heart Rate and Movement Monitoring.
Brief Title: A Home Telemonitoring System for Wearable Fetal-ECG and EHG Acquisition During Pregnancy
Acronym: AHTSWFEADP
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hao Li, Principal Investigator, Fudan University
Other Study IDs: PROFE23186I; 2022YFB4400800 (Other Grant/Funding Number: the National Key R&D Program of China)
Record Dates: First submitted 2023-08-29; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Uterine Contractions; Prolonged; Fetal Heart Rate or Rhythm Abnormality Affecting Fetus; Pregnancy Related; Home Range
Keywords: FECG; EHG
MeSH Terms: conditions — Homing Behavior

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: use wearable devices to monitoring fetal health conditions. — We used wearable devices and clinical cardiotocography (CTG) equipment to monitor pregnant women for 30 minutes to demonstrate the reliability of wearable devices.
  Other Names: Non-invasive monitoring; FECG; EHG

SUMMARY:
The goal of this observational is to compare in describing fetal health conditions. The main questions it aims to answer are:

* fetal electrocardiogram (fetal heart rate and fetal rhythm)
* electrohysterography (uterine contractions).

Participants will wear wearable devices and CTG equipment for monitoring for 30 minutes.If there is a comparison group: Researchers will compare clinical CTG equipment to see if this wearable device.

DETAILED DESCRIPTION:
The investigators put the patch of the wearable device on the abdomen of the pregnant woman and continued the test for thirty minutes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a gestational cycle greater than 36 weeks

Exclusion Criteria:

* male
* Pregnant women with a gestational cycle less than 36 weeks

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A wearable and remote fetal monitoring system is specifically developed for home use. It aims to overcome the limitations of conventional cardiotocography (CTG) devices by providing great user comfort and long-term continuous monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2023-08-06 (Actual)

PRIMARY OUTCOMES:
The performance of this system in extracting fetal electrocardiogram (FECG) | 2022.01-2023.08
  extract fetal QRS intervals and numbers from FECG
The performance of this system in extracting electrohysterography (EHG) | 2022.01-2023.08
  use the contractions consistency index (CCI) parameters to analyze the relation between our measured EHG signal and the UC signal recorded by clinical CTG equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Tingting Li, master, Principal Investigator — Fudan University
Locations (1):
- FetaCare, Shanghai, Pudong New District， Shanghai, China

IPD SHARING:
Plan to Share IPD: No